CLINICAL TRIAL: NCT04530344
Title: A Double-Blind, Vehicle-Controlled, Randomized Withdrawal and Treatment Extension Study to Assess the Long-Term Efficacy and Safety of Ruxolitinib Cream in Participants With Vitiligo
Brief Title: Assess the Long Term Efficacy and Safety of Ruxolitinib Cream in Participants With Vitiligo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCB 18424-308; 2020-000987-53 (EudraCT Number)
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Results first posted 2023-07-19 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Vitiligo
Keywords: INCB018424
MeSH Terms: conditions — Vitiligo | interventions — ruxolitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A : ruxolitinib cream (Experimental): Participants who achieve complete or almost complete facial repigmentation (achieve ≥ F VASI90) at Week 52 in the parent study will be assigned to Cohort A and will be randomized 1:1 to ruxolitinib cream.
  Interventions: Drug: ruxolitinib
- Cohort A : Vehicle (Placebo Comparator): Participants who achieve complete or almost complete facial repigmentation (ie, achieve ≥ F VASI90) at Week 52 in the parent study will be assigned to Cohort A and will be randomized 1:1 to vehicle cream.
  Interventions: Drug: Vehicle
- Cohort B : roxolitinib cream (Experimental): Participants who did not achieve ≥ F-VASI90 at Week 52 of the parent studies will be assigned to Cohort B and will continue ruxolitinib cream.
  Interventions: Drug: ruxolitinib

INTERVENTIONS:
Drug: ruxolitinib — ruxolitinib cream is a topical formulation applied as a thin film to affected areas BID.
  Other Names: INCB018424 Cream
  Arms: Cohort A : ruxolitinib cream; Cohort B : roxolitinib cream
Drug: Vehicle — Vehicle cream is a topical formulation applied as a thin film to affected areas.
  Arms: Cohort A : Vehicle

SUMMARY:
The purpose of this study is to evaluate the duration of response following withdrawal of ruxolitinib cream (Cohort A vehicle group), safety and maintenance of response with continued use of ruxolitinib cream in participants who have completed either Study NCT04052425 or NCT04057573 (parent studies) in which the participants will have been using ruxolitinib cream BID for the previous 28 to 52 weeks depending on their initial randomization in the parent study.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled and receiving treatment in INCB 18424-306 (NCT04052425) or INCB 18424-307 (NCT04057573) studies evaluating ruxolitinib cream in participants with vitiligo.
* Currently tolerating ruxolitinib cream in the parent study and no safety concerns per investigators judgment.
* Has demonstrated compliance, as assessed by the investigator, with the parent study protocol requirements.
* Willingness and ability to comply with scheduled visits, treatment plans, and any other study procedures indicated in this protocol.
* Male and female participants must be willing to take appropriate contraceptive measures to avoid pregnancy or fathering a child.
* Ability to comprehend and willingness to sign an ICF or written informed consent of the parent(s) or legal guardian and written assent from the participant when possible.

Exclusion Criteria:

* Has been permanently discontinued from study treatment in the parent study for any reason.
* Participants with an uncontrolled intercurrent illness or any concurrent condition that, in the investigator's opinion, would jeopardize the safety of the participant or compliance with the Protocol.
* Pregnant or breastfeeding woman.
* Participants who live with anyone participating in any current Incyte-sponsored ruxolitinib cream study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Butler, MD, Study Chair — Incyte Corporation
Locations (84):
- United States (44):
  - Cahaba Dermatology, Hoover, Alabama
  - Desert Sky Dermatology, Gilbert, Arizona
  - First Oc Dermatology, Fountain Valley, California
  - Center For Dermatology Cosmetic and Laser Surgery, Fremont, California
  - Marvel Clinical Research Llc, Huntington Beach, California
  - Vitiligo & Pigmentation Institute of Southern California, Los Angeles, California
  - Dermatology Research Associates, Los Angeles, California
  - Acrc Studies, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Colorado Medical Research Center Inc, Denver, Colorado
  - Harmony Medical Research Institute, Hialeah, Florida
  - Advanced Pharma, Miami, Florida
  - San Marcus Research Clinic Inc., Miami Lakes, Florida
  - Leavitt Medical Associates of Florida, Ormond Beach, Florida
  - Avita Clinical Research, Tampa, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Forcare Clinical Research Fcr Forward Clinical Trials, Inc, Tampa, Florida
  - Metabolic Research Institute Inc, West Palm Beach, Florida
  - Northwestern University, Chicago, Illinois
  - Randall Dermatology, West Lafayette, Indiana
  - Delricht Clinical Research - Clinedge - Ppds Baton Rouge, Baton Rouge, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Metro Boston Clinical Partners, Brighton, Massachusetts
  - Great Lakes Research Group Inc, Bay City, Michigan
  - Henry Ford Medical Center, Detroit, Michigan
  - Minnesota Clinical Study Center, Minneapolis, Minnesota
  - Jdr Dermatology Research, Las Vegas, Nevada
  - Suny Downstate Medical Center, Brooklyn, New York
  - Forest Hills Dermatology Group, Kew Gardens, New York
  - The Dermatology Specialists Greenwich, New York, New York
  - Icahn School of Medicine At Mount Sinai, New York, New York
  - Derm Research Center of New York Inc, Stony Brook, New York
  - Wake Research Associates Llc, Raleigh, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Central Sooner Research, Norman, Oklahoma
  - Kgl Skin Study Center, Broomall, Pennsylvania
  - Dermatology Associates of Plymouth Meeting, Plymouth Meeting, Pennsylvania
  - Palmetto Clinical Trial Services, Anderson, South Carolina
  - International Clinical Research Tennessee Llc, Murfreesboro, Tennessee
  - Innovative Dermatology, Plano, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - The Dermatology and Laser Center of San Antonio, San Antonio, Texas
  - Clinical Research Partners Llc, Richmond, Virginia
  - Dermatology Specialists of Spokane, Spokane, Washington
- Bulgaria (5):
  - Medical Center Unimed Eood, Sevlievo
  - Diagnostic Consultative Center Ii Sofia Eood, Sofia
  - University Multiprofile Hospital For Active Treatment Aleksandrovska, Sofia
  - Diagnostic Consultative Center Xxviii - Sofia - Eood, Sofia
  - Medical Center Eurohealth, Sofia
- Canada (8):
  - Dermatology Research Institute, Calgary, Alberta
  - Simcoderm Medical and Surgical Dermatology Center, Barrie, Ontario
  - Kingsway Clinical Research, Etobicoke, Ontario
  - Lynderm Research Inc, Markham, Ontario
  - Skin Centre For Dermatology, Peterborough, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - Xlr8 Medical Research, Windsor, Ontario
  - Siena Medical Research Corporation, Westmount, Quebec
- France (5):
  - Le Bateau Blanc, Martigues
  - Hopital Archet 2 Derm Dept, Nice
  - Centre Hospitalier Universitaire de Bordeaux - Hospital Haut-Leveque, Pessac
  - Hopital Charles Nicolle Chu Rouen Hospital de Bois-Guillaume, Rouen
  - Chu de Toulouse Hopital Larrey Centre de Reference Des Maladies Rares de La Peau Service de Dermatol, Toulouse
- Germany (4):
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - Hautarztpraxis Mahlow, Mahlow
  - Universitatsmedizin Der Johannes Gutenberg-Universitat Mainz Iii, Mainz
  - Universitatsklinik Munster Dermatologie, Münster
- Amsterdam University Medical Centre, Amsterdam, Netherlands
- Poland (14):
  - Synexus - Polska Sp Z Oo Oddzial W Gdansk, Gdansk
  - Synexus Polska Sp. Z O.O. Oddzial W Gdyni, Gdynia
  - Synexus - Sp Z Oo Oddzial W Katowice, Katowice
  - Synexus Affiliate - Krakowskie Centrum Medyczne, Krakow
  - Synexus Polska Sp Z Oo Oddzial W Lodzi, Lodz
  - Synexus Polska Sp Z Oo Oddzial W Czestochowie, Lublin
  - Dermedic Dr. Zdybski, Ostrowiec Świętokrzyski
  - Synexus Polska Sp. Z O.O. Oddzial W Poznaniu, Poznan
  - Lubeskie Centrum Diagnostyczne, Świdnik
  - Poradnia Dermatologiczno-Wenerologiczna Mediderm S.C. Nzoz, Torun
  - Synexus Polska Sp. Z O.O. Oddzial Warszawie, Warsaw
  - High-Med Przychodnia Specjalistycza, Warsaw
  - Synexus Polska Sp. Z O.O. Oddzial We Wroclawiu, Wroclaw
  - Dermmedica Sp. Z O.O., Wroclaw
- Spain (3):
  - Ico Hospital Germans Trias I Pujol, Badalona
  - Dermomedic, Madrid
  - Clinica Universidad de Navarra (Cun), Pamplona

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- [Derived] Rosmarin D, Pandya AG, Passeron T, Forman SB, Zdybski J, Amster M, Feser C, Papp KA, Nuara A, Kornacki D, Wei S, Ren H, Harris JE, Ezzedine K. Long-Term Integrated Safety Summary of Ruxolitinib Cream in Phase 3 Clinical Trials of Patients with Vitiligo. Dermatol Ther (Heidelb). 2025 Dec;15(12):3703-3716. doi: 10.1007/s13555-025-01555-3. Epub 2025 Oct 22. PMID 41125994

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 87 study centers in North America and Europe.
Pre-assignment Details: This randomized withdrawal and treatment-extension study (extension of treatment received in 2 parent studies: NCT04052425 or NCT04057573) was comprised of a 52-week extension treatment period and a 4-week safety follow-up period, starting 4 weeks (30 days) after the last application of study treatment or the last study visit.
Groups:
- Cohort A: Vehicle Cream BID: Participants who completed treatment and achieved ≥90% improvement from Baseline in the Facial Vitiligo Area Scoring Index score (≥F-VASI90) at Week 52 in either of 2 parent studies (NCT04052425 or NCT04057573). In this study, these participants were randomized to receive vehicle cream twice daily (BID) for 52 weeks. Participants who experienced relapse (<75% improvement from Baseline in the F-VASI score [<F-VASI75]) received open-label ruxolitinib 1.5% cream BID for the duration of the study.
- Cohort A: Ruxolitinib 1.5% Cream BID: Participants who completed treatment and achieved ≥F-VASI90 at Week 52 in either of 2 parent studies (NCT04052425 or NCT04057573). In this study, these participants were randomized to receive ruxolitinib 1.5% cream BID for 52 weeks. Participants who experienced relapse (<F-VASI75) received open-label ruxolitinib 1.5% cream BID for the duration of the study.
- Cohort B: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID: Participants who completed treatment (vehicle cream BID for 24 weeks and ruxolitinib 1.5% BID for 28 weeks) and did not achieve ≥F-VASI90 at Week 52 in either of 2 parent studies (NCT04052425 or NCT04057573). In this study, these participants applied ruxolitinib 1.5% cream BID for 52 weeks.
- Cohort B: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID: Participants who completed treatment (ruxolitinib 1.5% BID for 52 weeks) and did not achieve ≥F-VASI90 at Week 52 in either of 2 parent studies (NCT04052425 or NCT04057573). In this study, these participants applied ruxolitinib 1.5% cream BID for 52 weeks.
Period: Overall Study
Arm/Group | Cohort A: Vehicle Cream BID | Cohort A: Ruxolitinib 1.5% Cream BID | Cohort B: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Cohort B: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Started | 58 | 58 | 118 | 224
Completed | 41 | 50 | 92 | 173
Not Completed | 17 | 8 | 26 | 51
Not completed — Lost to Follow-up | 3 | 3 | 3 | 10
Not completed — Withdrawal by Subject | 14 | 5 | 18 | 33
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 1
Not completed — Pregnancy | 0 | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Site Closed Due to Noncompliance | 0 | 0 | 0 | 1
Not completed — Discontinued due to COVID-19 Pandemic | 0 | 0 | 1 | 0
Not completed — Missed Safety Follow-up Visit | 0 | 0 | 1 | 0
Not completed — Personal Reasons | 0 | 0 | 0 | 1
Not completed — Not Compliant with Protocol-specific Visit Window | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Vehicle Cream BID | Cohort A: Ruxolitinib 1.5% Cream BID | Cohort B: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Cohort B: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID | Total
Number analyzed (Participants) | 58 | 58 | 118 | 224 | 458
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (12.49) | 42.9 (15.95) | 39.7 (14.62) | 39.3 (16.45) | 39.9 (15.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 61 | 129 | 254
  Male | 27 | 25 | 57 | 95 | 204
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 3 | 3 | 8 | 18
  Black or African American | 5 | 4 | 3 | 11 | 23
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1 | 2
  Not Reported | 2 | 1 | 3 | 13 | 19
  White | 42 | 48 | 107 | 180 | 377
  Captured as Latino in Database | 1 | 0 | 0 | 0 | 1
  Persian | 1 | 0 | 0 | 0 | 1
  Indo-Caribbean | 1 | 0 | 0 | 0 | 1
  Jordanian | 1 | 0 | 0 | 0 | 1
  Brazilian | 0 | 1 | 0 | 0 | 1
  Guyana | 0 | 1 | 0 | 0 | 1
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Cape Verdean | 0 | 0 | 1 | 1 | 2
  Dominican Republic | 0 | 0 | 1 | 0 | 1
  Captured as Hispanic or Latino in Database | 0 | 0 | 0 | 1 | 1
  Iranian | 0 | 0 | 0 | 1 | 1
  Indian | 0 | 0 | 0 | 1 | 1
  North African | 0 | 0 | 0 | 1 | 1
  Middle Eastern | 0 | 0 | 0 | 1 | 1
  Arab//North-African | 0 | 0 | 0 | 1 | 1
  White/Black/Asian | 0 | 0 | 0 | 1 | 1
  Mexican | 0 | 0 | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 13 | 16 | 53 | 93
  Not Hispanic or Latino | 45 | 43 | 99 | 157 | 344
  Not Reported | 2 | 1 | 3 | 11 | 17
  Unknown | 0 | 0 | 0 | 1 | 1
  Captured as Other in Database | 0 | 1 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Time to Relapse (Defined as <F-VASI75)
Description: Relapse was defined as a loss of 75% improvement from Baseline in the Face Vitiligo Area Scoring Index score (F-VASI75) response, assessed as percentage improvement in the F-VASI score at Baseline (Day 1 of the parent study) to <75%.
Time Frame: from Week 52 (first visit of this Treatment Extension study) to Week 104 (end of treatment in this Treatment Extension study)
Population: Intent-to-Treat Long-term Extension (ITT-Ext) Population: randomized participants who achieved ≥90% improvement from Baseline in the F-VASI score (≥F-VASI90) at Week 52. Treatment groups were defined according to the treatment assignment at randomization regardless of the actual study medication the participant received. Week 52 was the first visit of this Treatment Extension study (visits were named to reflect continuation from the parent studies). Only participants in Cohort A were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cohort A: Vehicle Cream BID | Cohort A: Ruxolitinib 1.5% Cream BID | Cohort B: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Cohort B: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 56 | 55 | 0 | 0
days | NA [238.0 to NA] — The median and the upper limit of the confidence interval were not estimable because there were too few events of loss of F-VASI75 response. | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because there were too few events of loss of F-VASI75 response. |  |
Statistical Analysis 1: Comparison: Cohort A: Vehicle Cream BID vs Cohort A: Ruxolitinib 1.5% Cream BID; Cox regression model stratified by stratification factor (treatment assignment in the parent studies) was conducted to compare the difference in hazard rate between treatment and vehicle; Test type: Superiority; p = 0.0414, Log Rank; The p-value was based on the log-rank test stratified by randomization stratification factor between treatment and vehicle; Hazard Ratio (HR) = 0.422, 95% CI 2-sided [0.180 to 0.990]

2. Secondary Outcome: Time to Loss of Adequate Response
Description: Loss of adequate response was defined as a loss of 90% improvement from Baseline in the F-VASI score (F-VASI90) response, assessed as percentage improvement in the F-VASI score at Baseline (Day 1 of the parent study) to <90%.
Time Frame: as for outcome 1
Population: ITT-Ext Population. Week 52 was the first visit of this Treatment Extension study (visits were named to reflect continuation from the parent studies). Only participants in Cohort A were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cohort A: Vehicle Cream BID | Cohort A: Ruxolitinib 1.5% Cream BID | Cohort B: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Cohort B: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 56 | 55 | 0 | 0
days | 195.0 [113.0 to 372.0] | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because there were too few events of loss of F-VASI90 response. |  |
Statistical Analysis 1: Comparison: Cohort A: Vehicle Cream BID vs Cohort A: Ruxolitinib 1.5% Cream BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0003, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.316, 95% CI 2-sided [0.165 to 0.606]

3. Secondary Outcome: Percentage of Participants Achieving a ≥50% Improvement From Baseline in the Face Vitiligo Area Scoring Index (F-VASI50) Score During the Extension Treatment Period
Description: An F-VASI50 responder achieved at least 50% improvement from Baseline in F-VASI, measured by the percentage of vitiligo involvement (percentage of body surface area [BSA]) and the degree of depigmentation: 0% (no depigmentation), 10% (only specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), or 100% (no pigment). The percentage of BSA (hand unit) vitiligo involvement was estimated to the nearest 0.1% by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate the percentage of BSA vitiligo involvement. F-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site on the face and summing the values of all sites (possible range: 0-3; lower scores indicate increased improvement).
Time Frame: up to Week 104 of Treatment Extension (Week 52 was the first visit of this Treatment Extension study.)
Population: Full Analysis Set (FAS) without non-compliant site: all participants who received at least 1 dose of study drug at or after Week 52 (Baseline of Treatment Extension study). For participants who experienced relapse (<F-VASI75) and received open-label rescue treatment, only results before receiving open-label rescue treatment have been included. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Vehicle Cream BID | Cohort A: Ruxolitinib 1.5% Cream BID | Cohort B: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Cohort B: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 57 | 57 | 118 | 222
percentage of participants
  Week 52: number analyzed (Participants) | 57 | 57 | 118 | 221
  Week 52 | 98.2 [90.6 to 100.0] | 98.2 [90.6 to 100.0] | 45.8 [36.6 to 55.2] | 65.6 [58.9 to 71.9]
  Week 56: number analyzed (Participants) | 56 | 55 | 108 | 216
  Week 56 | 98.2 [90.4 to 100.0] | 96.4 [87.5 to 99.6] | 50.0 [40.2 to 59.8] | 69.4 [62.8 to 75.5]
  Week 60: number analyzed (Participants) | 48 | 52 | 107 | 211
  Week 60 | 97.9 [88.9 to 99.9] | 98.1 [89.7 to 100.0] | 54.2 [44.3 to 63.9] | 69.2 [62.5 to 75.4]
  Week 64: number analyzed (Participants) | 43 | 45 | 108 | 207
  Week 64 | 97.7 [87.7 to 99.9] | 100.0 [92.1 to 100.0] | 58.3 [48.5 to 67.7] | 72.0 [65.3 to 78.0]
  Week 68: number analyzed (Participants) | 41 | 45 | 107 | 210
  Week 68 | 95.1 [83.5 to 99.4] | 100.0 [92.1 to 100.0] | 63.6 [53.7 to 72.6] | 77.1 [70.9 to 82.6]
  Week 80: number analyzed (Participants) | 30 | 45 | 99 | 194
  Week 80 | 96.7 [82.8 to 99.9] | 100.0 [92.1 to 100.0] | 65.7 [55.4 to 74.9] | 78.9 [72.4 to 84.4]
  Week 92: number analyzed (Participants) | 23 | 43 | 94 | 179
  Week 92 | 100.0 [85.2 to 100.0] | 97.7 [87.7 to 99.9] | 66.0 [55.5 to 75.4] | 84.4 [78.2 to 89.3]
  Week 104: number analyzed (Participants) | 23 | 38 | 93 | 177
  Week 104 | 95.7 [78.1 to 99.9] | 100.0 [90.7 to 100.0] | 69.9 [59.5 to 79.0] | 86.4 [80.5 to 91.1]

4. Secondary Outcome: Percentage of Participants Achieving a ≥75% Improvement From Baseline in the F-VASI (F-VASI75) Score During the Extension Treatment Period
Description: An F-VASI75 responder achieved at least 75% improvement from Baseline in F-VASI, measured by the percentage of vitiligo involvement (percentage of BSA) and the degree of depigmentation: 0% (no depigmentation), 10% (only specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), or 100% (no pigment). The percentage of BSA (hand unit) vitiligo involvement was estimated to the nearest 0.1% by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate the percentage of BSA vitiligo involvement. F-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site on the face and summing the values of all sites (possible range: 0-3; lower scores indicate increased improvement).
Time Frame: up to Week 104 of Treatment Extension (Week 52 was the first visit of this Treatment Extension study.)
Population: FAS without non-compliant site. For participants who experienced relapse (<F-VASI75) and received open-label rescue treatment, only results before receiving open-label rescue treatment have been included. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Vehicle Cream BID | Cohort A: Ruxolitinib 1.5% Cream BID | Cohort B: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Cohort B: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 57 | 57 | 118 | 222
percentage of participants
  Week 52: number analyzed (Participants) | 57 | 57 | 118 | 221
  Week 52 | 98.2 [90.6 to 100.0] | 98.2 [90.6 to 100.0] | 16.1 [10.0 to 24.0] | 30.8 [24.8 to 37.3]
  Week 56: number analyzed (Participants) | 56 | 55 | 108 | 216
  Week 56 | 96.4 [87.7 to 99.6] | 96.4 [87.5 to 99.6] | 23.1 [15.6 to 32.2] | 34.7 [28.4 to 41.5]
  Week 60: number analyzed (Participants) | 48 | 52 | 107 | 211
  Week 60 | 95.8 [85.7 to 99.5] | 90.4 [79.0 to 96.8] | 29.0 [20.6 to 38.5] | 40.8 [34.1 to 47.7]
  Week 64: number analyzed (Participants) | 43 | 45 | 108 | 207
  Week 64 | 95.3 [84.2 to 99.4] | 97.8 [88.2 to 99.9] | 30.6 [22.1 to 40.2] | 43.5 [36.6 to 50.5]
  Week 68: number analyzed (Participants) | 41 | 45 | 107 | 210
  Week 68 | 87.8 [73.8 to 95.9] | 100.0 [92.1 to 100.0] | 34.6 [25.6 to 44.4] | 48.6 [41.6 to 55.5]
  Week 80: number analyzed (Participants) | 30 | 45 | 99 | 194
  Week 80 | 90.0 [73.5 to 97.9] | 100.0 [92.1 to 100.0] | 43.4 [33.5 to 53.8] | 54.6 [47.4 to 61.8]
  Week 92: number analyzed (Participants) | 23 | 43 | 94 | 179
  Week 92 | 100.0 [85.2 to 100.0] | 97.7 [87.7 to 99.9] | 47.9 [37.5 to 58.4] | 60.3 [52.8 to 67.6]
  Week 104: number analyzed (Participants) | 23 | 38 | 93 | 177
  Week 104 | 95.7 [78.1 to 99.9] | 97.4 [86.2 to 99.9] | 47.3 [36.9 to 57.9] | 66.1 [58.6 to 73.0]

5. Secondary Outcome: Percentage of Participants Achieving a ≥90% Improvement From Baseline in the F-VASI (F-VASI90) Score During the Extension Treatment Period
Description: An F-VASI90 responder achieved at least 90% improvement from Baseline in F-VASI, measured by the percentage of vitiligo involvement (percentage of BSA) and the degree of depigmentation: 0% (no depigmentation), 10% (only specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), or 100% (no pigment). The percentage of BSA (hand unit) vitiligo involvement was estimated to the nearest 0.1% by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate the percentage of BSA vitiligo involvement. F-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site on the face and summing the values of all sites (possible range: 0-3; lower scores indicate increased improvement).
Time Frame: up to Week 104 of Treatment Extension (Week 52 was the first visit of this Treatment Extension study.)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Vehicle Cream BID | Cohort A: Ruxolitinib 1.5% Cream BID | Cohort B: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Cohort B: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 57 | 57 | 118 | 222
percentage of participants
  Week 52: number analyzed (Participants) | 57 | 57 | 118 | 221
  Week 52 | 98.2 [90.6 to 100.0] | 96.5 [87.9 to 99.6] | 0.0 [0.0 to 3.1] | 2.3 [0.7 to 5.2]
  Week 56: number analyzed (Participants) | 56 | 55 | 108 | 216
  Week 56 | 89.3 [78.1 to 96.0] | 94.5 [84.9 to 98.9] | 3.7 [1.0 to 9.2] | 8.3 [5.0 to 12.9]
  Week 60: number analyzed (Participants) | 48 | 52 | 107 | 211
  Week 60 | 83.3 [69.8 to 92.5] | 86.5 [74.2 to 94.4] | 8.4 [3.9 to 15.4] | 15.2 [10.6 to 20.7]
  Week 64: number analyzed (Participants) | 43 | 45 | 108 | 207
  Week 64 | 72.1 [56.3 to 84.7] | 93.3 [81.7 to 98.6] | 11.1 [5.9 to 18.6] | 15.5 [10.8 to 21.1]
  Week 68: number analyzed (Participants) | 41 | 45 | 107 | 210
  Week 68 | 68.3 [51.9 to 81.9] | 95.6 [84.9 to 99.5] | 12.1 [6.6 to 19.9] | 22.4 [16.9 to 28.6]
  Week 80: number analyzed (Participants) | 30 | 45 | 99 | 194
  Week 80 | 80.0 [61.4 to 92.3] | 97.8 [88.2 to 99.9] | 22.2 [14.5 to 31.7] | 30.4 [24.0 to 37.4]
  Week 92: number analyzed (Participants) | 23 | 43 | 94 | 179
  Week 92 | 78.3 [56.3 to 92.5] | 93.0 [80.9 to 98.5] | 24.5 [16.2 to 34.4] | 32.4 [25.6 to 39.8]
  Week 104: number analyzed (Participants) | 23 | 38 | 93 | 177
  Week 104 | 69.6 [47.1 to 86.8] | 92.1 [78.6 to 98.3] | 28.0 [19.1 to 38.2] | 33.9 [27.0 to 41.4]

6. Secondary Outcome: Mean F-VASI Scores During the Extension Treatment Period
Description: F-VASI was measured by the percentage of vitiligo involvement (percentage of BSA) and the degree of depigmentation: 0% (no depigmentation), 10% (only specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), or 100% (no pigment). The percentage of BSA (hand unit) vitiligo involvement was estimated to the nearest 0.1% by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate the percentage of BSA vitiligo involvement. F-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site on the face and summing the values of all sites (possible range: 0-3; lower scores indicate increased improvement).
Time Frame: up to Week 104 of Treatment Extension (Week 52 was the first visit of this Treatment Extension study.)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cohort A: Vehicle Cream BID | Cohort A: Ruxolitinib 1.5% Cream BID | Cohort B: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Cohort B: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 57 | 57 | 118 | 222
scores on a scale
  Baseline | 0.86 (0.492) | 0.99 (0.644) | 0.88 (0.543) | 0.91 (0.550)
  Week 52: number analyzed (Participants) | 57 | 57 | 118 | 221
  Week 52 | 0.05 (0.110) | 0.07 (0.181) | 0.51 (0.459) | 0.39 (0.374)
  Week 56: number analyzed (Participants) | 56 | 55 | 108 | 216
  Week 56 | 0.05 (0.108) | 0.07 (0.186) | 0.50 (0.475) | 0.38 (0.372)
  Week 60: number analyzed (Participants) | 48 | 52 | 107 | 211
  Week 60 | 0.06 (0.145) | 0.09 (0.186) | 0.45 (0.450) | 0.35 (0.375)
  Week 64: number analyzed (Participants) | 43 | 45 | 108 | 207
  Week 64 | 0.08 (0.131) | 0.08 (0.230) | 0.43 (0.456) | 0.33 (0.350)
  Week 68: number analyzed (Participants) | 41 | 45 | 107 | 210
  Week 68 | 0.11 (0.199) | 0.04 (0.081) | 0.40 (0.430) | 0.31 (0.352)
  Week 80: number analyzed (Participants) | 30 | 45 | 99 | 194
  Week 80 | 0.05 (0.082) | 0.04 (0.108) | 0.36 (0.426) | 0.27 (0.345)
  Week 92: number analyzed (Participants) | 23 | 43 | 94 | 179
  Week 92 | 0.04 (0.055) | 0.04 (0.076) | 0.38 (0.471) | 0.23 (0.281)
  Week 104: number analyzed (Participants) | 23 | 38 | 93 | 177
  Week 104 | 0.06 (0.109) | 0.04 (0.083) | 0.37 (0.493) | 0.21 (0.280)

7. Secondary Outcome: Change From Baseline in F-VASI Scores During the Extension Treatment Period
Description: F-VASI was measured by the percentage of vitiligo involvement (percentage of BSA) and the degree of depigmentation: 0% (no depigmentation), 10% (only specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), or 100% (no pigment). The percentage of BSA (hand unit) vitiligo involvement was estimated to the nearest 0.1% by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate the percentage of BSA vitiligo involvement. F-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site on the face and summing the values of all sites (possible range: 0-3; lower scores indicate increased improvement). Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; up to Week 104 of Treatment Extension (Week 52 was the first visit of this Treatment Extension study.)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cohort A: Vehicle Cream BID | Cohort A: Ruxolitinib 1.5% Cream BID | Cohort B: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Cohort B: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 57 | 57 | 118 | 222
scores on a scale
  Week 52: number analyzed (Participants) | 57 | 57 | 118 | 221
  Week 52 | -0.81 (0.464) | -0.92 (0.591) | -0.37 (0.346) | -0.51 (0.448)
  Week 56: number analyzed (Participants) | 56 | 55 | 108 | 216
  Week 56 | -0.82 (0.492) | -0.90 (0.594) | -0.39 (0.370) | -0.54 (0.457)
  Week 60: number analyzed (Participants) | 48 | 52 | 107 | 211
  Week 60 | -0.84 (0.447) | -0.87 (0.570) | -0.43 (0.402) | -0.55 (0.457)
  Week 64: number analyzed (Participants) | 43 | 45 | 108 | 207
  Week 64 | -0.80 (0.442) | -0.87 (0.527) | -0.44 (0.423) | -0.58 (0.452)
  Week 68: number analyzed (Participants) | 41 | 45 | 107 | 210
  Week 68 | -0.73 (0.316) | -0.86 (0.518) | -0.46 (0.437) | -0.61 (0.476)
  Week 80: number analyzed (Participants) | 30 | 45 | 99 | 194
  Week 80 | -0.75 (0.360) | -0.86 (0.508) | -0.49 (0.471) | -0.64 (0.478)
  Week 92: number analyzed (Participants) | 23 | 43 | 94 | 179
  Week 92 | -0.76 (0.341) | -0.87 (0.548) | -0.48 (0.531) | -0.69 (0.488)
  Week 104: number analyzed (Participants) | 23 | 38 | 93 | 177
  Week 104 | -0.72 (0.380) | -0.92 (0.561) | -0.50 (0.557) | -0.68 (0.514)

8. Secondary Outcome: Percent Change From Baseline in F-VASI Scores During the Extension Treatment Period
Description: F-VASI was measured by the percentage of vitiligo involvement (percentage of BSA) and the degree of depigmentation: 0% (no depigmentation), 10% (only specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), or 100% (no pigment). The percentage of BSA (hand unit) vitiligo involvement was estimated to the nearest 0.1% by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate the percentage of BSA vitiligo involvement. F-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site on the face and summing the values of all sites (possible range: 0-3; lower scores indicate increased improvement). Percentage change = ([post-BL value minus BL value]/BL value) X 100.
Time Frame: Baseline (BL); up to Week 104 of Treatment Extension (Week 52 was the first visit of this Treatment Extension study.)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Cohort A: Vehicle Cream BID | Cohort A: Ruxolitinib 1.5% Cream BID | Cohort B: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Cohort B: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 57 | 57 | 118 | 222
percentage change
  Week 52: number analyzed (Participants) | 57 | 57 | 118 | 221
  Week 52 | -94.45 (14.069) | -94.50 (8.990) | -44.32 (27.775) | -54.72 (31.006)
  Week 56: number analyzed (Participants) | 56 | 55 | 108 | 216
  Week 56 | -93.79 (14.981) | -93.21 (12.573) | -46.19 (30.728) | -57.38 (31.256)
  Week 60: number analyzed (Participants) | 48 | 52 | 107 | 211
  Week 60 | -93.85 (9.087) | -92.04 (13.198) | -50.55 (30.537) | -60.17 (30.147)
  Week 64: number analyzed (Participants) | 43 | 45 | 108 | 207
  Week 64 | -89.64 (23.562) | -94.87 (8.079) | -52.32 (32.826) | -62.94 (27.427)
  Week 68: number analyzed (Participants) | 41 | 45 | 107 | 210
  Week 68 | -87.98 (19.644) | -96.25 (4.633) | -55.27 (32.433) | -65.55 (30.388)
  Week 80: number analyzed (Participants) | 30 | 45 | 99 | 194
  Week 80 | -93.24 (13.062) | -96.65 (4.683) | -58.60 (34.839) | -69.38 (29.091)
  Week 92: number analyzed (Participants) | 23 | 43 | 94 | 179
  Week 92 | -95.77 (5.586) | -94.95 (10.366) | -55.44 (49.855) | -73.77 (25.490)
  Week 104: number analyzed (Participants) | 23 | 38 | 93 | 177
  Week 104 | -90.53 (17.763) | -95.86 (7.213) | -56.53 (57.087) | -73.84 (31.780)

9. Secondary Outcome: Percentage of Participants Achieving a ≥50% Improvement From Baseline in the Total Body Vitiligo Area Scoring Index (T-VASI50) Score During the Extension Treatment Period
Description: A T-VASI50 responder achieved at least 50% improvement from Baseline in T-VASI, calculated with contributions from 6 sites. The percentage of vitiligo involvement was estimated in hand units (percentage of BSA estimated to nearest 0.1%) by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate percent BSA vitiligo involvement. The degree of depigmentation for each site was estimated to the nearest percentage: 0% (no depigmentation present), 10% (only specks of depigmentation present), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment present), 100% (no pigment present). T-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site and summing the values (range: 0-100; lower scores indicate increased improvement).
Time Frame: up to Week 104 of Treatment Extension (Week 52 was the first visit of this Treatment Extension study.)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Vehicle Cream BID | Cohort A: Ruxolitinib 1.5% Cream BID | Cohort B: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Cohort B: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 57 | 57 | 118 | 222
percentage of participants
  Week 52: number analyzed (Participants) | 57 | 57 | 118 | 221
  Week 52 | 80.7 [68.1 to 90.0] | 71.9 [58.5 to 83.0] | 16.9 [10.7 to 25.0] | 42.5 [35.9 to 49.3]
  Week 56: number analyzed (Participants) | 56 | 55 | 108 | 216
  Week 56 | 76.8 [63.6 to 87.0] | 72.7 [59.0 to 83.9] | 16.7 [10.2 to 25.1] | 45.8 [39.1 to 52.7]
  Week 60: number analyzed (Participants) | 48 | 52 | 107 | 211
  Week 60 | 83.3 [69.8 to 92.5] | 75.0 [61.1 to 86.0] | 19.6 [12.6 to 28.4] | 49.8 [42.8 to 56.7]
  Week 64: number analyzed (Participants) | 43 | 45 | 108 | 207
  Week 64 | 74.4 [58.8 to 86.5] | 82.2 [67.9 to 92.0] | 21.3 [14.0 to 30.2] | 50.7 [43.7 to 57.7]
  Week 68: number analyzed (Participants) | 41 | 45 | 107 | 210
  Week 68 | 70.7 [54.5 to 83.9] | 84.4 [70.5 to 93.5] | 29.9 [21.4 to 39.5] | 54.3 [47.3 to 61.2]
  Week 80: number analyzed (Participants) | 30 | 45 | 99 | 194
  Week 80 | 80.0 [61.4 to 92.3] | 86.7 [73.2 to 94.9] | 39.4 [29.7 to 49.7] | 57.7 [50.4 to 64.8]
  Week 92: number analyzed (Participants) | 23 | 43 | 94 | 179
  Week 92 | 73.9 [51.6 to 89.8] | 86.0 [72.1 to 94.7] | 48.9 [38.5 to 59.5] | 61.5 [53.9 to 68.6]
  Week 104: number analyzed (Participants) | 23 | 38 | 93 | 177
  Week 104 | 60.9 [38.5 to 80.3] | 89.5 [75.2 to 97.1] | 54.8 [44.2 to 65.2] | 63.8 [56.3 to 70.9]

10. Secondary Outcome: Percentage of Participants Achieving a ≥75% Improvement From Baseline in the T-VASI (T-VASI75) Score During the Extension Treatment Period
Description: A T-VASI75 responder achieved at least 75% improvement from Baseline in T-VASI, calculated with contributions from 6 sites. The percentage of vitiligo involvement was estimated in hand units (percentage of BSA estimated to nearest 0.1%) by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate percent BSA vitiligo involvement. The degree of depigmentation for each site was estimated to the nearest percentage: 0% (no depigmentation present), 10% (only specks of depigmentation present), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment present), 100% (no pigment present). T-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site and summing the values (range: 0-100; lower scores indicate increased improvement).
Time Frame: up to Week 104 of Treatment Extension (Week 52 was the first visit of this Treatment Extension study.)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Vehicle Cream BID | Cohort A: Ruxolitinib 1.5% Cream BID | Cohort B: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Cohort B: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 57 | 57 | 118 | 222
percentage of participants
  Week 52: number analyzed (Participants) | 57 | 57 | 118 | 221
  Week 52 | 38.6 [26.0 to 52.4] | 42.1 [29.1 to 55.9] | 3.4 [0.9 to 8.5] | 12.2 [8.2 to 17.3]
  Week 56: number analyzed (Participants) | 56 | 55 | 108 | 216
  Week 56 | 42.9 [29.7 to 56.8] | 43.6 [30.3 to 57.7] | 4.6 [1.5 to 10.5] | 13.4 [9.2 to 18.7]
  Week 60: number analyzed (Participants) | 48 | 52 | 107 | 211
  Week 60 | 45.8 [31.4 to 60.8] | 38.5 [25.3 to 53.0] | 4.7 [1.5 to 10.6] | 14.2 [9.8 to 19.7]
  Week 64: number analyzed (Participants) | 43 | 45 | 108 | 207
  Week 64 | 39.5 [25.0 to 55.6] | 48.9 [33.7 to 64.2] | 3.7 [1.0 to 9.2] | 16.9 [12.1 to 22.7]
  Week 68: number analyzed (Participants) | 41 | 45 | 107 | 210
  Week 68 | 39.0 [24.2 to 55.5] | 42.2 [27.7 to 57.8] | 6.5 [2.7 to 13.0] | 22.4 [16.9 to 28.6]
  Week 80: number analyzed (Participants) | 30 | 45 | 99 | 194
  Week 80 | 53.3 [34.3 to 71.7] | 48.9 [33.7 to 64.2] | 10.1 [5.0 to 17.8] | 23.7 [17.9 to 30.3]
  Week 92: number analyzed (Participants) | 23 | 43 | 94 | 179
  Week 92 | 43.5 [23.2 to 65.5] | 53.5 [37.7 to 68.8] | 12.8 [6.8 to 21.2] | 29.1 [22.5 to 36.3]
  Week 104: number analyzed (Participants) | 23 | 38 | 93 | 177
  Week 104 | 39.1 [19.7 to 61.5] | 55.3 [38.3 to 71.4] | 18.3 [11.0 to 27.6] | 30.5 [23.8 to 37.9]

11. Secondary Outcome: Percentage of Participants Achieving a ≥90% Improvement From Baseline in the T-VASI (T-VASI90) Score During the Extension Treatment Period
Description: A T-VASI90 responder achieved at least 90% improvement from Baseline in T-VASI, calculated with contributions from 6 sites. The percentage of vitiligo involvement was estimated in hand units (percentage of BSA estimated to nearest 0.1%) by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate percent BSA vitiligo involvement. The degree of depigmentation for each site was estimated to the nearest percentage: 0% (no depigmentation present), 10% (only specks of depigmentation present), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment present), 100% (no pigment present). T-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site and summing the values (range: 0-100; lower scores indicate increased improvement).
Time Frame: up to Week 104 of Treatment Extension (Week 52 was the first visit of this Treatment Extension study.)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Vehicle Cream BID | Cohort A: Ruxolitinib 1.5% Cream BID | Cohort B: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Cohort B: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 57 | 57 | 118 | 222
percentage of participants
  Week 52: number analyzed (Participants) | 57 | 57 | 118 | 221
  Week 52 | 12.3 [5.1 to 23.7] | 12.3 [5.1 to 23.7] | 0.0 [0.0 to 3.1] | 2.3 [0.7 to 5.2]
  Week 56: number analyzed (Participants) | 56 | 55 | 108 | 216
  Week 56 | 12.5 [5.2 to 24.1] | 14.5 [6.5 to 26.7] | 0.0 [0.0 to 3.4] | 3.2 [1.3 to 6.6]
  Week 60: number analyzed (Participants) | 48 | 52 | 107 | 211
  Week 60 | 16.7 [7.5 to 30.2] | 17.3 [8.2 to 30.3] | 0.0 [0.0 to 3.4] | 3.8 [1.7 to 7.3]
  Week 64: number analyzed (Participants) | 43 | 45 | 108 | 207
  Week 64 | 20.9 [10.0 to 36.0] | 20.0 [9.6 to 34.6] | 0.0 [0.0 to 3.4] | 2.9 [1.1 to 6.2]
  Week 68: number analyzed (Participants) | 41 | 45 | 107 | 210
  Week 68 | 22.0 [10.6 to 37.6] | 20.0 [9.6 to 34.6] | 0.9 [0.0 to 5.1] | 4.3 [2.0 to 8.0]
  Week 80: number analyzed (Participants) | 30 | 45 | 99 | 194
  Week 80 | 20.0 [7.7 to 38.6] | 20.0 [9.6 to 34.6] | 1.0 [0.0 to 5.5] | 6.7 [3.6 to 11.2]
  Week 92: number analyzed (Participants) | 23 | 43 | 94 | 179
  Week 92 | 21.7 [7.5 to 43.7] | 20.9 [10.0 to 36.0] | 2.1 [0.3 to 7.5] | 8.9 [5.2 to 14.1]
  Week 104: number analyzed (Participants) | 23 | 38 | 93 | 177
  Week 104 | 21.7 [7.5 to 43.7] | 23.7 [11.4 to 40.2] | 3.2 [0.7 to 9.1] | 9.6 [5.7 to 14.9]

12. Secondary Outcome: Mean T-VASI Scores During the Extension Treatment Period
Description: T-VASI was calculated with contributions from 6 sites. The percentage of vitiligo involvement was estimated in hand units (percentage of BSA estimated to nearest 0.1%) by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate percent BSA vitiligo involvement. The degree of depigmentation for each site was estimated to the nearest percentage: 0% (no depigmentation present), 10% (only specks of depigmentation present), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment present), 100% (no pigment present). T-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site and summing the values (range: 0-100; lower scores indicate increased improvement).
Time Frame: up to Week 104 of Treatment Extension (Week 52 was the first visit of this Treatment Extension study.)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cohort A: Vehicle Cream BID | Cohort A: Ruxolitinib 1.5% Cream BID | Cohort B: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Cohort B: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 57 | 57 | 118 | 222
scores on a scale
  Baseline | 6.06 (2.056) | 6.27 (2.030) | 6.69 (2.150) | 6.74 (2.006)
  Week 52: number analyzed (Participants) | 57 | 57 | 118 | 221
  Week 52 | 2.38 (2.206) | 2.36 (1.805) | 5.25 (3.248) | 3.90 (2.132)
  Week 56: number analyzed (Participants) | 56 | 55 | 108 | 216
  Week 56 | 2.39 (2.253) | 2.31 (1.843) | 5.06 (3.151) | 3.80 (2.213)
  Week 60: number analyzed (Participants) | 48 | 52 | 107 | 211
  Week 60 | 2.21 (2.176) | 2.30 (1.841) | 4.86 (3.150) | 3.58 (2.122)
  Week 64: number analyzed (Participants) | 43 | 45 | 108 | 207
  Week 64 | 2.33 (2.210) | 1.94 (1.717) | 4.85 (3.317) | 3.57 (2.051)
  Week 68: number analyzed (Participants) | 41 | 45 | 107 | 210
  Week 68 | 2.45 (2.231) | 1.76 (1.378) | 4.51 (3.060) | 3.43 (2.160)
  Week 80: number analyzed (Participants) | 30 | 45 | 99 | 194
  Week 80 | 2.05 (2.233) | 1.73 (1.331) | 4.18 (3.036) | 3.18 (2.017)
  Week 92: number analyzed (Participants) | 23 | 43 | 94 | 179
  Week 92 | 2.17 (1.913) | 1.65 (1.244) | 4.12 (3.477) | 3.04 (2.128)
  Week 104: number analyzed (Participants) | 23 | 38 | 93 | 177
  Week 104 | 2.86 (3.269) | 1.54 (1.227) | 4.00 (4.208) | 2.92 (2.061)

13. Secondary Outcome: Change From Baseline in T-VASI Scores During the Extension Treatment Period
Description: T-VASI was calculated with contributions from 6 sites. The percentage of vitiligo involvement was estimated in hand units (percentage of BSA estimated to nearest 0.1%) by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate percent BSA vitiligo involvement. The degree of depigmentation for each site was estimated to the nearest percentage: 0% (no depigmentation present), 10% (only specks of depigmentation present), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment present), 100% (no pigment present). T-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site and summing the values (range: 0-100; lower scores indicate increased improvement). Change from Baseline=post-Baseline value minus the Baseline value.
Time Frame: Baseline; up to Week 104 of Treatment Extension (Week 52 was the first visit of this Treatment Extension study.)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cohort A: Vehicle Cream BID | Cohort A: Ruxolitinib 1.5% Cream BID | Cohort B: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Cohort B: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 57 | 57 | 118 | 222
scores on a scale
  Week 52: number analyzed (Participants) | 57 | 57 | 118 | 221
  Week 52 | -3.68 (1.564) | -3.91 (1.526) | -1.45 (2.271) | -2.83 (1.938)
  Week 56: number analyzed (Participants) | 56 | 55 | 108 | 216
  Week 56 | -3.71 (1.615) | -3.91 (1.503) | -1.69 (2.217) | -2.97 (2.086)
  Week 60: number analyzed (Participants) | 48 | 52 | 107 | 211
  Week 60 | -3.79 (1.692) | -3.95 (1.585) | -1.83 (2.161) | -3.16 (2.027)
  Week 64: number analyzed (Participants) | 43 | 45 | 108 | 207
  Week 64 | -3.60 (2.033) | -4.20 (1.569) | -1.84 (2.375) | -3.21 (2.060)
  Week 68: number analyzed (Participants) | 41 | 45 | 107 | 210
  Week 68 | -3.44 (1.789) | -4.24 (1.534) | -2.21 (2.273) | -3.35 (2.143)
  Week 80: number analyzed (Participants) | 30 | 45 | 99 | 194
  Week 80 | -3.79 (1.663) | -4.26 (1.519) | -2.49 (2.175) | -3.55 (2.109)
  Week 92: number analyzed (Participants) | 23 | 43 | 94 | 179
  Week 92 | -3.85 (1.545) | -4.33 (1.673) | -2.61 (2.624) | -3.73 (2.246)
  Week 104: number analyzed (Participants) | 23 | 38 | 93 | 177
  Week 104 | -3.05 (2.156) | -4.48 (1.702) | -2.71 (3.479) | -3.84 (2.151)

14. Secondary Outcome: Percent Change From Baseline in T-VASI Scores During the Extension Treatment Period
Description: T-VASI was calculated with contributions from 6 sites. The percentage of vitiligo involvement was estimated in hand units (percentage of BSA estimated to nearest 0.1%) by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate percent BSA vitiligo involvement. The degree of depigmentation for each site was estimated to the nearest percentage: 0% (no depigmentation present), 10% (only specks of depigmentation present), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment present), 100% (no pigment present). T-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site and summing the values (range: 0-100; lower scores indicate increased improvement). Percentage change = ([post-BL value minus BL value]/BL value) X 100.
Time Frame: Baseline; up to Week 104 of Treatment Extension (Week 52 was the first visit of this Treatment Extension study.)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Cohort A: Vehicle Cream BID | Cohort A: Ruxolitinib 1.5% Cream BID | Cohort B: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Cohort B: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 57 | 57 | 118 | 222
percentage change
  Week 52: number analyzed (Participants) | 57 | 57 | 118 | 221
  Week 52 | -65.01 (23.969) | -64.95 (21.547) | -24.75 (2.271) | -42.14 (25.783)
  Week 56: number analyzed (Participants) | 56 | 55 | 108 | 216
  Week 56 | -65.16 (24.916) | -65.69 (22.042) | -28.05 (30.487) | -43.91 (27.408)
  Week 60: number analyzed (Participants) | 48 | 52 | 107 | 211
  Week 60 | -66.83 (26.478) | -65.58 (22.910) | -31.01 (28.944) | -47.00 (26.089)
  Week 64: number analyzed (Participants) | 43 | 45 | 108 | 207
  Week 64 | -62.82 (33.328) | -70.44 (20.212) | -30.85 (32.898) | -46.96 (26.395)
  Week 68: number analyzed (Participants) | 41 | 45 | 107 | 210
  Week 68 | -61.40 (29.204) | -71.89 (17.942) | -35.53 (32.135) | -49.41 (27.629)
  Week 80: number analyzed (Participants) | 30 | 45 | 99 | 194
  Week 80 | -68.99 (26.870) | -72.21 (17.852) | -40.97 (30.033) | -52.48 (26.991)
  Week 92: number analyzed (Participants) | 23 | 43 | 94 | 179
  Week 92 | -66.95 (24.885) | -72.55 (19.152) | -43.34 (34.425) | -55.00 (28.995)
  Week 104: number analyzed (Participants) | 23 | 38 | 93 | 177
  Week 104 | -58.38 (35.533) | -74.66 (17.727) | -45.52 (41.968) | -56.96 (27.409)

15. Secondary Outcome: Mean Facial Body Surface Area (F-BSA) During the Extension Treatment Period
Description: F-BSA involvement was the proportion of the facial body surface area with vitiligo. The area "Face" was defined as including the area on the forehead to the original hairline, on the cheek to the jawline vertically to the jawline and laterally from the corner of the mouth to the tragus. The area "Face" did not include surface area of the lips, scalp, ears, or neck, but included the nose and eyelids. Body surface area assessment was performed by the Palmar Method. Body surface area was estimated to the nearest 0.1%. The approximate size of the participant's entire palmar surface (i.e., the palm plus 5 digits) was considered as 1% BSA, and the approximate size of the participant's thumb was considered as 0.1% BSA. Data are presented as the percentage of BSA involvement in the face as compared to total BSA.
Time Frame: up to Week 104 of Treatment Extension (Week 52 was the first visit of this Treatment Extension study.)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage BSA
Arm/Group | Cohort A: Vehicle Cream BID | Cohort A: Ruxolitinib 1.5% Cream BID | Cohort B: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Cohort B: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 57 | 57 | 118 | 222
percentage BSA
  Baseline | 0.92 (0.498) | 1.10 (0.745) | 1.01 (0.632) | 1.02 (0.636)
  Week 52: number analyzed (Participants) | 57 | 57 | 118 | 221
  Week 52 | 0.18 (0.240) | 0.27 (0.401) | 0.81 (0.641) | 0.70 (0.568)
  Week 56: number analyzed (Participants) | 56 | 55 | 108 | 216
  Week 56 | 0.18 (0.198) | 0.27 (0.416) | 0.77 (0.638) | 0.67 (0.572)
  Week 60: number analyzed (Participants) | 48 | 51 | 107 | 211
  Week 60 | 0.20 (0.225) | 0.25 (0.309) | 0.73 (0.616) | 0.63 (0.557)
  Week 64: number analyzed (Participants) | 43 | 45 | 108 | 207
  Week 64 | 0.20 (0.206) | 0.20 (0.271) | 0.71 (0.607) | 0.61 (0.566)
  Week 68: number analyzed (Participants) | 41 | 45 | 107 | 210
  Week 68 | 0.22 (0.258) | 0.16 (0.183) | 0.67 (0.581) | 0.57 (0.548)
  Week 80: number analyzed (Participants) | 30 | 45 | 99 | 194
  Week 80 | 0.12 (0.138) | 0.15 (0.200) | 0.62 (0.565) | 0.55 (0.564)
  Week 92: number analyzed (Participants) | 23 | 43 | 94 | 179
  Week 92 | 0.10 (0.130) | 0.15 (0.180) | 0.64 (0.595) | 0.49 (0.527)
  Week 104: number analyzed (Participants) | 23 | 38 | 93 | 177
  Week 104 | 0.13 (0.154) | 0.15 (0.181) | 0.62 (0.602) | 0.47 (0.509)

16. Secondary Outcome: Change From Baseline in F-BSA During the Extension Treatment Period
Description: F-BSA involvement was the proportion of the facial body surface area with vitiligo. The area "Face" was defined as including the area on the forehead to the original hairline, on the cheek to the jawline vertically to the jawline and laterally from the corner of the mouth to the tragus. The area "Face" did not include surface area of the lips, scalp, ears, or neck, but included the nose and eyelids. Body surface area assessment was performed by the Palmar Method. Body surface area was estimated to the nearest 0.1%. The approximate size of the participant's entire palmar surface (i.e., the palm plus 5 digits) was considered as 1% BSA, and the approximate size of the participant's thumb was considered as 0.1% BSA. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Data are presented as the percentage of BSA involvement in the face as compared to total BSA.
Time Frame: Baseline; up to Week 104 of Treatment Extension (Week 52 was the first visit of this Treatment Extension study.)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage BSA
Arm/Group | Cohort A: Vehicle Cream BID | Cohort A: Ruxolitinib 1.5% Cream BID | Cohort B: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Cohort B: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 57 | 57 | 118 | 222
percentage BSA
  Week 52: number analyzed (Participants) | 57 | 57 | 118 | 221
  Week 52 | -0.74 (0.402) | -0.83 (0.638) | -0.20 (0.313) | -0.31 (0.435)
  Week 56: number analyzed (Participants) | 56 | 55 | 108 | 216
  Week 56 | -0.76 (0.458) | -0.82 (0.672) | -0.25 (0.345) | -0.35 (0.433)
  Week 60: number analyzed (Participants) | 48 | 51 | 107 | 211
  Week 60 | -0.77 (0.441) | -0.80 (0.601) | -0.28 (0.364) | -0.38 (0.454)
  Week 64: number analyzed (Participants) | 43 | 45 | 108 | 207
  Week 64 | -0.74 (0.446) | -0.83 (0.625) | -0.29 (0.417) | -0.41 (0.457)
  Week 68: number analyzed (Participants) | 41 | 45 | 107 | 210
  Week 68 | -0.69 (0.345) | -0.86 (0.657) | -0.31 (0.425) | -0.45 (0.489)
  Week 80: number analyzed (Participants) | 30 | 45 | 99 | 194
  Week 80 | -0.74 (0.381) | -0.87 (0.637) | -0.37 (0.494) | -0.48 (0.521)
  Week 92: number analyzed (Participants) | 23 | 43 | 94 | 179
  Week 92 | -0.76 (0.374) | -0.87 (0.678) | -0.36 (0.558) | -0.54 (0.532)
  Week 104: number analyzed (Participants) | 23 | 38 | 93 | 177
  Week 104 | -0.70 (0.400) | -0.93 (0.716) | -0.39 (0.604) | -0.54 (0.548)

17. Secondary Outcome: Percent Change From Baseline in F-BSA During the Extension Treatment Period
Description: F-BSA involvement was the proportion of the facial body surface area with vitiligo. The area "Face" was defined as including the area on the forehead to the original hairline, on the cheek to the jawline vertically to the jawline and laterally from the corner of the mouth to the tragus. The area "Face" did not include surface area of the lips, scalp, ears, or neck, but included the nose and eyelids. Body surface area assessment was performed by the Palmar Method. Body surface area was estimated to the nearest 0.1%. The approximate size of the participant's entire palmar surface (i.e., the palm plus 5 digits) was considered as 1% BSA, and the approximate size of the participant's thumb was considered as 0.1% BSA. Percentage change = ([post-Baseline (BL) value minus BL value]/BL value) X 100.
Time Frame: Baseline; up to Week 104 of Treatment Extension (Week 52 was the first visit of this Treatment Extension study.)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Cohort A: Vehicle Cream BID | Cohort A: Ruxolitinib 1.5% Cream BID | Cohort B: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Cohort B: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 57 | 57 | 118 | 222
percentage change
  Week 52: number analyzed (Participants) | 57 | 57 | 118 | 221
  Week 52 | -80.75 (18.726) | -76.75 (23.470) | -22.15 (28.268) | -29.06 (36.354)
  Week 56: number analyzed (Participants) | 56 | 55 | 108 | 216
  Week 56 | -80.23 (21.828) | -74.42 (35.048) | -26.20 (30.604) | -33.66 (33.944)
  Week 60: number analyzed (Participants) | 48 | 51 | 107 | 211
  Week 60 | -79.20 (19.463) | -77.67 (20.946) | -30.04 (30.751) | -36.86 (33.289)
  Week 64: number analyzed (Participants) | 43 | 45 | 108 | 207
  Week 64 | -75.92 (32.175) | -80.06 (22.142) | -30.67 (33.473) | -39.58 (31.992)
  Week 68: number analyzed (Participants) | 41 | 45 | 107 | 210
  Week 68 | -77.11 (23.565) | -83.14 (21.999) | -32.60 (34.575) | -43.61 (32.549)
  Week 80: number analyzed (Participants) | 30 | 45 | 99 | 194
  Week 80 | -84.55 (18.730) | -84.67 (22.014) | -36.79 (36.826) | -46.38 (34.407)
  Week 92: number analyzed (Participants) | 23 | 43 | 94 | 179
  Week 92 | -87.81 (15.738) | -83.24 (23.746) | -34.05 (50.762) | -51.96 (31.510)
  Week 104: number analyzed (Participants) | 23 | 38 | 93 | 177
  Week 104 | -82.87 (23.245) | -84.09 (22.920) | -35.82 (52.646) | -52.85 (32.983)

18. Secondary Outcome: Mean Total Body Surface Area (T-BSA) During the Extension Treatment Period
Description: T-BSA involvement was the proportion of the body surface area with vitiligo. Body surface area assessment was performed by the Palmar Method. Body surface area was estimated to the nearest 0.1%. The approximate size of the participant's entire palmar surface (i.e., the palm plus 5 digits) was considered as 1% BSA, and the approximate size of the participant's thumb was considered as 0.1% BSA. Data are presented as the percentage of BSA involvement in the total body.
Time Frame: up to Week 104 of Treatment Extension (Week 52 was the first visit of this Treatment Extension study.)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage BSA
Arm/Group | Cohort A: Vehicle Cream BID | Cohort A: Ruxolitinib 1.5% Cream BID | Cohort B: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Cohort B: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 57 | 57 | 118 | 222
percentage BSA
  Baseline | 6.79 (2.157) | 6.85 (1.924) | 7.42 (2.064) | 7.49 (2.006)
  Week 52: number analyzed (Participants) | 57 | 57 | 118 | 221
  Week 52 | 4.09 (2.838) | 4.20 (2.640) | 6.95 (3.403) | 5.96 (2.352)
  Week 56: number analyzed (Participants) | 56 | 55 | 108 | 216
  Week 56 | 4.11 (2.880) | 4.13 (2.788) | 6.73 (3.281) | 5.81 (2.558)
  Week 60: number analyzed (Participants) | 48 | 51 | 107 | 211
  Week 60 | 3.77 (2.756) | 4.09 (2.833) | 6.61 (3.262) | 5.64 (2.479)
  Week 64: number analyzed (Participants) | 43 | 45 | 108 | 207
  Week 64 | 3.98 (3.087) | 3.49 (2.452) | 6.67 (3.448) | 5.64 (2.483)
  Week 68: number analyzed (Participants) | 41 | 45 | 107 | 210
  Week 68 | 3.92 (2.813) | 3.27 (2.310) | 6.46 (3.239) | 5.51 (2.682)
  Week 80: number analyzed (Participants) | 30 | 45 | 99 | 194
  Week 80 | 3.72 (3.151) | 3.18 (2.232) | 6.09 (3.313) | 5.27 (2.581)
  Week 92: number analyzed (Participants) | 23 | 43 | 94 | 179
  Week 92 | 3.94 (2.834) | 3.04 (2.194) | 5.96 (3.646) | 5.15 (2.741)
  Week 104: number analyzed (Participants) | 23 | 38 | 93 | 177
  Week 104 | 4.56 (4.156) | 2.93 (2.301) | 5.91 (4.475) | 5.07 (2.699)

19. Secondary Outcome: Change From Baseline in T-BSA During the Extension Treatment Period
Description: T-BSA involvement was the proportion of the body surface area with vitiligo. Body surface area assessment was performed by the Palmar Method. Body surface area was estimated to the nearest 0.1%. The approximate size of the participant's entire palmar surface (i.e., the palm plus 5 digits) was considered as 1% BSA, and the approximate size of the participant's thumb was considered as 0.1% BSA. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Data are presented as the percentage of BSA involvement in the total body.
Time Frame: Baseline; up to Week 104 of Treatment Extension (Week 52 was the first visit of this Treatment Extension study.)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage BSA
Arm/Group | Cohort A: Vehicle Cream BID | Cohort A: Ruxolitinib 1.5% Cream BID | Cohort B: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Cohort B: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 57 | 57 | 118 | 222
percentage BSA
  Week 52: number analyzed (Participants) | 57 | 57 | 118 | 221
  Week 52 | -2.70 (1.830) | -2.64 (1.906) | -0.47 (2.325) | -1.52 (1.711)
  Week 56: number analyzed (Participants) | 56 | 55 | 108 | 216
  Week 56 | -2.74 (1.918) | -2.70 (1.983) | -0.73 (2.238) | -1.71 (2.059)
  Week 60: number analyzed (Participants) | 48 | 51 | 107 | 211
  Week 60 | -2.95 (1.910) | -2.75 (2.195) | -0.80 (2.128) | -1.86 (1.978)
  Week 64: number analyzed (Participants) | 43 | 45 | 108 | 207
  Week 64 | -2.73 (2.528) | -3.22 (1.883) | -0.73 (2.432) | -1.90 (2.052)
  Week 68: number analyzed (Participants) | 41 | 45 | 107 | 210
  Week 68 | -2.73 (1.958) | -3.34 (1.922) | -0.98 (2.262) | -2.03 (2.180)
  Week 80: number analyzed (Participants) | 30 | 45 | 99 | 194
  Week 80 | -3.05 (2.083) | -3.42 (1.809) | -1.31 (2.341) | -2.21 (2.169)
  Week 92: number analyzed (Participants) | 23 | 43 | 94 | 179
  Week 92 | -3.03 (1.664) | -3.58 (1.938) | -1.49 (2.753) | -2.36 (2.380)
  Week 104: number analyzed (Participants) | 23 | 38 | 93 | 177
  Week 104 | -2.18 (2.723) | -3.72 (2.075) | -1.52 (3.672) | -2.42 (2.307)

20. Secondary Outcome: Percent Change From Baseline in T-BSA During the Extension Treatment Period
Description: T-BSA involvement was the proportion of the body surface area with vitiligo. Body surface area assessment was performed by the Palmar Method. Body surface area was estimated to the nearest 0.1%. The approximate size of the participant's entire palmar surface (i.e., the palm plus 5 digits) was considered as 1% BSA, and the approximate size of the participant's thumb was considered as 0.1% BSA. Percentage change = ([post-Baseline (BL) value minus BL value]/BL value) X 100.
Time Frame: Baseline; up to Week 104 of Treatment Extension (Week 52 was the first visit of this Treatment Extension study.)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Cohort A: Vehicle Cream BID | Cohort A: Ruxolitinib 1.5% Cream BID | Cohort B: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Cohort B: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 57 | 57 | 118 | 222
percentage change
  Week 52: number analyzed (Participants) | 57 | 57 | 118 | 221
  Week 52 | -43.81 (27.916) | -41.50 (28.747) | -8.54 (28.806) | -20.57 (23.042)
  Week 56: number analyzed (Participants) | 56 | 55 | 108 | 216
  Week 56 | -44.22 (29.590) | -43.12 (29.489) | -11.96 (28.156) | -22.98 (26.032)
  Week 60: number analyzed (Participants) | 48 | 51 | 107 | 211
  Week 60 | -47.61 (29.237) | -43.09 (31.608) | -13.40 (26.410) | -25.12 (25.564)
  Week 64: number analyzed (Participants) | 43 | 45 | 108 | 207
  Week 64 | -43.29 (40.045) | -50.59 (27.166) | -12.00 (30.202) | -25.15 (26.860)
  Week 68: number analyzed (Participants) | 41 | 45 | 107 | 210
  Week 68 | -44.53 (30.086) | -52.51 (26.921) | -15.01 (29.093) | -27.59 (28.476)
  Week 80: number analyzed (Participants) | 30 | 45 | 99 | 194
  Week 80 | -50.51 (33.794) | -53.98 (25.682) | -20.22 (30.154) | -29.92 (27.996)
  Week 92: number analyzed (Participants) | 23 | 43 | 94 | 179
  Week 92 | -48.53 (29.457) | -55.56 (26.401) | -22.84 (33.708) | -31.98 (30.805)
  Week 104: number analyzed (Participants) | 23 | 38 | 93 | 177
  Week 104 | -40.84 (40.076) | -57.40 (27.898) | -24.26 (42.193) | -32.96 (29.907)

21. Secondary Outcome: Percentage of Participants Achieving a Vitiligo Noticeability Scale (VNS) Score of 4 or 5 During the Extension Treatment Period
Description: The VNS is a patient-reported measure of vitiligo treatment success that is rated on a 5-point scale. The Baseline facial photograph was shown to the participants for reference, and a mirror was provided for the participants to assess the vitiligo on their face. The participant was asked to respond to the following query: Compared with before treatment, how noticeable is the vitiligo now? Responses: (1) more noticeable, (2) as noticeable, (3) slightly less noticeable, (4) a lot less noticeable, and (5) no longer noticeable.
Time Frame: Baseline; up to Week 104 of Treatment Extension (Week 52 was the first visit of this Treatment Extension study.)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Vehicle Cream BID | Cohort A: Ruxolitinib 1.5% Cream BID | Cohort B: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Cohort B: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 57 | 57 | 118 | 222
percentage of participants
  Week 52: number analyzed (Participants) | 57 | 57 | 118 | 221
  Week 52 | 49.1 [35.6 to 62.7] | 42.1 [29.1 to 55.9] | 11.9 [6.6 to 19.1] | 35.3 [29.0 to 42.0]
  Week 56: number analyzed (Participants) | 56 | 55 | 108 | 216
  Week 56 | 48.2 [34.7 to 62.0] | 34.5 [22.2 to 48.6] | 20.4 [13.2 to 29.2] | 30.1 [24.1 to 36.7]
  Week 60: number analyzed (Participants) | 49 | 52 | 107 | 210
  Week 60 | 46.9 [32.5 to 61.7] | 28.8 [17.1 to 43.1] | 19.6 [12.6 to 28.4] | 27.6 [21.7 to 34.2]
  Week 64: number analyzed (Participants) | 43 | 45 | 108 | 206
  Week 64 | 53.5 [37.7 to 68.8] | 37.8 [23.8 to 53.5] | 23.1 [15.6 to 32.2] | 28.2 [22.1 to 34.8]
  Week 68: number analyzed (Participants) | 41 | 45 | 107 | 210
  Week 68 | 46.3 [30.7 to 62.6] | 46.7 [31.7 to 62.1] | 20.6 [13.4 to 29.5] | 33.8 [27.4 to 40.6]
  Week 80: number analyzed (Participants) | 31 | 45 | 99 | 195
  Week 80 | 38.7 [21.8 to 57.8] | 42.2 [27.7 to 57.8] | 28.3 [19.7 to 38.2] | 32.8 [26.3 to 39.9]
  Week 92: number analyzed (Participants) | 23 | 43 | 95 | 180
  Week 92 | 39.1 [19.7 to 61.5] | 37.2 [23.0 to 53.3] | 28.4 [19.6 to 38.6] | 41.1 [33.8 to 48.7]
  Week 104: number analyzed (Participants) | 23 | 38 | 93 | 178
  Week 104 | 56.5 [34.5 to 76.8] | 50.0 [33.4 to 66.6] | 30.1 [21.0 to 40.5] | 43.3 [35.9 to 50.9]

22. Secondary Outcome: Change From Week 52 in Dermatology Life Quality Index (DLQI) Total Score During the Extension Treatment Period
Description: The DLQI is a simple, 10-question validated questionnaire to measure how much the skin problem has affected the participant over the previous 7 days. Participants age ≥16 years answered the questionnaire with: (1) very much; (2) a lot; (3) a little; or (4) not at all. The questionnaire was analyzed under 6 headings: Symptoms and feelings (Questions 1 and 2); Daily activities (Questions 3 and 4); Leisure (Questions 5 and 6); Work and school (Question 7); Personal relations (Questions 8 and 9); and Treatment (Question 10). The scoring of each question is as follows: very much = 3; a lot = 2; a little = 1; not at all = 0; not relevant = 0. For Question 7, "prevented work or studying"=3. The total score ranges from 0 to 30; higher scores indicate higher quality of life. Change from Week 52 was calculated as the post-Week 52 value minus the Week 52 value.
Time Frame: Week 52; up to up to Week 104 of Extension Study (Week 52 was the first visit of this Treatment Extension study.)
Population: FAS without non-compliant site. For participants who experienced relapse (<F-VASI75) and received open-label rescue treatment, only results before receiving open-label rescue treatment have been included. Only participants who were ≥16 years old with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cohort A: Vehicle Cream BID | Cohort A: Ruxolitinib 1.5% Cream BID | Cohort B: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Cohort B: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 54 | 51 | 114 | 200
scores on a scale
  Week 52 | 2.87 (3.059) | 4.10 (4.784) | 3.69 (3.428) | 3.53 (4.150)
  Change from Week 52 at Week 56: number analyzed (Participants) | 53 | 49 | 104 | 194
  Change from Week 52 at Week 56 | 0.11 (2.054) | -0.47 (1.757) | -0.05 (2.138) | -0.22 (2.483)
  Change from Week 52 at Week 60: number analyzed (Participants) | 46 | 46 | 103 | 188
  Change from Week 52 at Week 60 | 0.37 (2.388) | 0.13 (2.227) | 0.28 (2.491) | 0.24 (2.929)
  Change from Week 52 at Week 64: number analyzed (Participants) | 40 | 40 | 104 | 184
  Change from Week 52 at Week 64 | 0.35 (2.578) | 0.18 (2.630) | -0.06 (2.712) | -0.14 (2.350)
  Change from Week 52 at Week 68: number analyzed (Participants) | 38 | 40 | 103 | 188
  Change from Week 52 at Week 68 | -0.08 (2.508) | -0.15 (2.202) | -0.17 (2.501) | 0.08 (2.454)
  Change from Week 52 at Week 80: number analyzed (Participants) | 29 | 40 | 95 | 175
  Change from Week 52 at Week 80 | 0.03 (3.006) | -0.23 (2.315) | -0.77 (2.871) | -0.13 (2.809)
  Change from Week 52 at Week 92: number analyzed (Participants) | 22 | 39 | 91 | 160
  Change from Week 52 at Week 92 | 0.27 (2.354) | -0.23 (1.898) | -0.89 (2.383) | -0.22 (2.941)
  Change from Week 52 at Week 104: number analyzed (Participants) | 21 | 35 | 89 | 158
  Change from Week 52 at Week 104 | 0.57 (2.135) | -0.40 (1.538) | -0.48 (2.277) | -0.06 (2.813)

23. Secondary Outcome: Change From Week 52 in Children's Dermatology Life Quality Index (CDLQI) Total Score During the Extension Treatment Period
Description: The CDLQI is the youth/children's version of the DLQI. The DLQI is a simple, 10-question validated questionnaire to measure how much the skin problem has affected the participant over the previous 7 days. Participants age <16 years answered the questionnaire with: (1) very much; (2) a lot; (3) a little; or (4) not at all. The questionnaire was analyzed under 6 headings: Symptoms and feelings (Questions 1 and 2); Leisure (Questions 4, 5, and 6); School or holidays (Question 7); Personal relationships (Questions 3 and 8); Sleep (Question 9); and Treatment (Question 10). The scoring of each question is as follows: very much = 3; quite a lot = 2; only a little = 1; not at all = 0; question unanswered = 0. The total score ranges from 0 to 30; higher scores indicate higher quality of life. Change from Week 52 was calculated as the post-Week 52 value minus the Week 52 value.
Time Frame: Week 52; up to Week 104 of Treatment Extension (Week 52 was the first visit of this Treatment Extension study.)
Population: FAS without non-compliant site. For participants who experienced relapse (<F-VASI75) and received open-label rescue treatment, only results before receiving open-label rescue treatment have been included. Only participants who were <16 years old with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cohort A: Vehicle Cream BID | Cohort A: Ruxolitinib 1.5% Cream BID | Cohort B: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Cohort B: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 3 | 6 | 4 | 22
scores on a scale
  Week 52 | 1.67 (2.887) | 1.00 (0.632) | 1.25 (1.893) | 2.32 (3.872)
  Change from Week 52 at Week 56 | -1.00 (2.646) | -0.17 (0.753) | 0.00 (0.816) | 0.36 (1.989)
  Change from Week 52 at Week 60 | 0.00 (0.000) | -0.50 (0.548) | -0.50 (0.577) | -0.41 (2.108)
  Change from Week 52 at Week 64: number analyzed (Participants) | 3 | 5 | 4 | 22
  Change from Week 52 at Week 64 | -1.33 (2.309) | 0.00 (0.707) | -1.00 (1.414) | -0.36 (1.399)
  Change from Week 52 at Week 68: number analyzed (Participants) | 3 | 5 | 4 | 22
  Change from Week 52 at Week 68 | -0.67 (1.155) | 0.40 (1.140) | 0.50 (0.577) | -0.23 (1.541)
  Change from Week 52 at Week 80: number analyzed (Participants) | 2 | 5 | 4 | 20
  Change from Week 52 at Week 80 | -2.00 (2.828) | -0.40 (0.548) | -0.75 (1.708) | 0.15 (1.814)
  Change from Week 52 at Week 92: number analyzed (Participants) | 1 | 4 | 4 | 20
  Change from Week 52 at Week 92 | NA (NA) — The mean and standard deviation cannot be calculated for a single participant. | 0.25 (1.258) | -0.25 (0.957) | 0.70 (3.614)
  Change from Week 52 at Week 104: number analyzed (Participants) | 2 | 3 | 4 | 20
  Change from Week 52 at Week 104 | -0.50 (0.707) | -0.67 (1.155) | -1.25 (1.893) | -0.20 (4.086)

24. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: A TEAE was defined as any adverse event (AE) reported for the first time or the worsening of a pre-existing event after the first application of study drug in this study. An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment.
Time Frame: up to approximately Week 108 (Week 52 was the first visit of this Treatment Extension study.)
Population: FAS
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID: Participants who completed treatment and achieved ≥90% improvement from Baseline in the Facial Vitiligo Area Scoring Index score (≥F-VASI90) at Week 52 in either of 2 parent studies (NCT04052425 or NCT04057573). In this study, these participants were randomized to receive vehicle cream twice daily (BID) for 52 weeks. These participants experienced relapse (<F-VASI75) and received open-label ruxolitinib 1.5% cream BID for the duration of the study.
Arm/Group | Cohort A: Vehicle Cream BID | Cohort A: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Cohort A: Ruxolitinib 1.5% Cream BID | Cohort B: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Cohort B: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 58 | 23 | 58 | 118 | 224
Participants | 21 | 3 | 32 | 59 | 114

25. Secondary Outcome: Trough Plasma Concentrations of Ruxolitinib at Week 80 and Week 104
Description: The steady-state plasma concentration was assessed. Pharmacokinetic blood samples could have been collected at any time prior to study drug application at the site at the Week 80 visit and at any time at the Week 104 (End of Trial) visit. Results from the two parent studies indicated that steady state was reached at or before Week 4, and that, hence, the use of vehicle or ruxolitinib 1.5% in the first 52 weeks of treatment had no impact on the ruxolitinib plasma concentration at the Week 80 and Week 104 (End of Treatment) visits. Thus, the two Cohort B cohorts were combined into a single arm for data analysis in this study.
Time Frame: Weeks 80 (predose); Week 104 (any time post-dose) (Week 52 was the first visit of this Treatment Extension study.)
Population: Pharmacokinetic (PK) Evaluable Population: all participants who received at least 1 dose of ruxolitinib cream and provided at least 1 measurable post-dose PK sample/assessment. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: nanomolar
Groups:
- Cohort B: Ruxolitinib 1.5% Cream BID: Participants who completed treatment (vehicle cream BID for 24 weeks and ruxolitinib 1.5% BID for 28 weeks or ruxolitinib 1.5% BID for 52 weeks) and did not achieve ≥F-VASI90 at Week 52 in either of 2 parent studies (NCT04052425 or NCT04057573). In this study, these participants applied ruxolitinib 1.5% cream BID for 52 weeks.
- Cohorts A and B: Ruxolitinib 1.5% Cream BID: Participants who completed treatment and achieved ≥F-VASI90 at Week 52 in either of 2 parent studies (NCT04052425 or NCT04057573). Participants who completed treatment (vehicle cream BID for 24 weeks and ruxolitinib 1.5% BID for 28 weeks or ruxolitinib 1.5% BID for 52 weeks) and did not achieve ≥F-VASI90 at Week 52 in either of 2 parent studies (NCT04052425 or NCT04057573). In this study, these participants (58 from Cohort A; 289 from Cohort B) applied ruxolitinib 1.5% cream BID for 52 weeks.
Arm/Group | Cohort A: Ruxolitinib 1.5% Cream BID | Cohort B: Ruxolitinib 1.5% Cream BID | Cohorts A and B: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 54 | 293 | 347
nanomolar
  12 to <18 years: number analyzed (Participants) | 8 | 40 | 48
  12 to <18 years | 7.28 (11.7) | 5.56 (10.5) | 5.85 (10.6)
  18 to <65 years: number analyzed (Participants) | 43 | 229 | 272
  18 to <65 years | 15.1 (19.5) | 12.7 (17.2) | 13.1 (17.6)
  ≥65 years: number analyzed (Participants) | 3 | 24 | 27
  ≥65 years | 13.0 (9.44) | 25.7 (20.9) | 24.3 (20.2)
  Overall | 13.8 (18.1) | 12.8 (17.4) | 12.9 (17.5)

ADVERSE EVENTS:
Time Frame: up to approximately Week 108 (Week 52 was the first visit of this Treatment Extension study.)
Description: Treatment-emergent adverse events, defined as adverse events reported for the first time or the worsening of pre-existing events after the first application of study drug, have been reported.
Groups:
- Vehicle Cream BID: Participants who completed treatment and achieved ≥90% improvement from Baseline in the Facial Vitiligo Area Scoring Index score (≥F-VASI90) at Week 52 in either of 2 parent studies (NCT04052425 or NCT04057573). In this study, these participants were randomized to receive vehicle cream twice daily (BID) for 52 weeks. Participants who experienced relapse (<75% improvement from Baseline in the F-VASI score [<F-VASI75]) received open-label ruxolitinib 1.5% cream BID for the duration of the study.
- Ruxolitinib 1.5% Cream BID: Participants who completed treatment and achieved ≥F-VASI90 at Week 52 in either of 2 parent studies (NCT04052425 or NCT04057573). In this study, these participants were randomized to receive ruxolitinib 1.5% cream BID for 52 weeks, or were randomized to receive vehicle cream BID but experienced relapse (<F-VASI75) and received open-label ruxolitinib 1.5% cream BID for the duration of the study. Participants who completed treatment (vehicle cream BID for 24 weeks and ruxolitinib 1.5% BID for 28 weeks) and did not achieve ≥F-VASI90 at Week 52 in either of 2 parent studies (NCT04052425 or NCT04057573). In this study, these participants applied ruxolitinib 1.5% cream BID for 52 weeks. Participants who completed treatment (ruxolitinib 1.5% BID for 52 weeks) and did not achieve ≥F-VASI90 at Week 52 in either of 2 parent studies (NCT04052425 or NCT04057573). In this study, these participants applied ruxolitinib 1.5% cream BID for 52 weeks.
- Total: Total
Arm/Group | Vehicle Cream BID | Ruxolitinib 1.5% Cream BID | Total
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/423 | 0/458
Serious Adverse Events (participants affected / at risk) | 0/58 | 12/423 | 12/458
Other Adverse Events (participants affected / at risk) | 6/58 | 55/423 | 61/458
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Cream BID (N=58) | Ruxolitinib 1.5% Cream BID (N=423) | Total (N=458)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Otosclerosis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Pelvic prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Rectocele (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (2)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Cream BID (N=58) | Ruxolitinib 1.5% Cream BID (N=423) | Total (N=458)
COVID-19 (Infections and infestations) | 6 (6) | 55 (57) | 61 (63)

LIMITATIONS AND CAVEATS:
Data from participants at a single site (N = 2) were removed from all efficacy analyses performed on the ITT-Ext Population and FAS Cohort A owing to noncompliance with the Protocol in the parent study resulting in serious concerns with data quality.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/44/NCT04530344/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/44/NCT04530344/SAP_001.pdf